CLINICAL TRIAL: NCT02943447
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, and Efficacy of GS-9674 in Subjects With Primary Biliary Cholangitis Without Cirrhosis
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of Cilofexor in Adults With Primary Biliary Cholangitis Without Cirrhosis
Acronym: PBC-Phase 2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated because of the availability of alternate therapies for primary biliary cholangitis (PBC).
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-427-4024; 2016-002443-42 (EudraCT Number)
Record Dates: First submitted 2016-06-13; First posted 2016-10-24 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — cilofexor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cilofexor 30 mg (Blinded Study Phase) (Experimental): Cilofexor 30 mg + placebo to match cilofexor 100 mg for 12 weeks.
  Interventions: Drug: Cilofexor; Drug: Placebo to match cilofexor
- Cilofexor 100 mg (Blinded Study Phase) (Experimental): Cilofexor 100 mg + placebo to match cilofexor 30 mg for 12 weeks.
  Interventions: Drug: Cilofexor; Drug: Placebo to match cilofexor
- Placebo (Blinded Study Phase) (Placebo Comparator): Placebo to match cilofexor 30 mg + placebo to match cilofexor 100 mg for 12 weeks.
  Interventions: Drug: Placebo to match cilofexor
- Cilofexor (Open Label Extension Phase) (Experimental): Following the Blinded Study Phase, eligible participants may have the option to receive open-label cilofexor 100 mg for an additional 96 weeks.
  Interventions: Drug: Cilofexor

INTERVENTIONS:
Drug: Cilofexor — Tablet(s) administered orally once daily, with food
  Other Names: GS-9674
  Arms: Cilofexor (Open Label Extension Phase); Cilofexor 100 mg (Blinded Study Phase); Cilofexor 30 mg (Blinded Study Phase)
Drug: Placebo to match cilofexor — Tablet(s) administered orally once daily, with food
  Arms: Cilofexor 100 mg (Blinded Study Phase); Cilofexor 30 mg (Blinded Study Phase); Placebo (Blinded Study Phase)

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of cilofexor in adults with primary biliary cholangitis (PBC).

ELIGIBILITY:
Key Inclusion Criteria:

* Meets all of the following conditions

  * Definite or probable PBC as defined by at least 2 of the 3 following criteria:

    * Serum alkaline phosphatase (ALP) > the upper limit of normal (ULN)
    * Presence of anti-mitochondrial antibodies (AMA) in serum (≥ 1:40 on immunofluorescence)
    * Liver histological findings consistent with PBC including nonsuppurative, destructive cholangitis affecting mainly the interlobular bile and septal bile ducts
  * Serum ALP > 1.67 x ULN and/or total bilirubin >ULN but ≤ 2 x ULN
  * Ursodeoxycholic acid (UDCA) use at a stable dose for at least 12 months or intolerant of UDCA with no UDCA use for at least 12 months before screening
* Screening FibroSURE/FibroTest® < 0.75 unless a historical liver biopsy within 12 months of screening does not reveal cirrhosis. In adults with Gilbert's syndrome or hemolysis, FibroSURE/FibroTest will be calculated using direct bilirubin instead of total bilirubin.

Key Exclusion Criteria:

* Alanine aminotransferase (ALT) > 5 x ULN
* Total bilirubin > 2 x ULN
* International normalized ratio (INR) > 1.2 unless on anticoagulant therapy
* Other causes of liver disease including viral, metabolic, alcoholic, and other autoimmune conditions. Participants with hepatic steatosis may be included if there is no evidence of nonalcoholic steatohepatitis (NASH) in the opinion of the investigator or on liver biopsy.
* Use of fibrates or obeticholic acid within 3 months prior to screening through the end of treatment
* Cirrhosis of the liver as defined by any of the following:

  * Historical liver biopsy demonstrating cirrhosis (eg, Ludwig stage 4 or Ishak stage ≥ 5)
  * History of decompensated liver disease, including ascites, hepatic encephalopathy or variceal bleeding
  * Liver stiffness > 16.9 kPa by FibroScan®

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (22):
- United States (12):
  - Sacramento, California
  - Aurora, Colorado
  - Lakewood Rch, Florida
  - Miami, Florida
  - Marietta, Georgia
  - Saint Paul, Minnesota
  - Arlington, Texas
  - Dallas, Texas
  - Houston, Texas
  - Charlottesville, Virginia
  - Newport News, Virginia
  - Seattle, Washington
- Austria (2):
  - Graz, Styria
  - Vienna, Vienna
- Canada (5):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Toronto, Ontario
  - Vaughan, Ontario
- United Kingdom (3):
  - Birmingham, England
  - London, England
  - Norwich, England

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kowdley KV, Minuk GY, Pagadala MR, Gulamhusein A, Swain MG, Neff GW, et al. The Nonsteroidal Farnesoid X Receptor (FXR) Agonist Cilofexor Improves Liver Biochemistry in Patients with Primary Biliary Cholangitis (PBC): A Phase 2, Randomized, Placebo-Controlled Trial [Abstract 45]. Hepatology AASLD Abstracts 2019;70 (Suppl 1):31A-2A.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States, Canada, United Kingdom, and Austria. The first participant was screened on 01 December 2016. The last study visit occurred on 4 September 2019.
Pre-assignment Details: 130 participants were screened.
Groups:
- Cilofexor 100 mg: Blinded Study Phase: Cilofexor 100 mg tablet + placebo to match cilofexor 30 mg tablet orally once daily for 12 weeks.
  Open-Label Extension (OLE) Phase: Following Blinded Study Phase, participants willing to enter OLE Phase received open-label cilofexor 100 mg tablet orally once daily for 97.4 weeks.
- Cilofexor 30 mg: Blinded Study Phase: Cilofexor 30 mg tablet + placebo to match cilofexor 100 mg tablet orally once daily for 12 weeks.
  OLE Phase: Following Blinded Study Phase, participants willing to enter OLE Phase received open-label cilofexor 100 mg tablet orally once daily for 96.1 weeks.
- Placebo: Blinded Study Phase: Placebo to match cilofexor 100 mg tablet + placebo to match cilofexor 30 mg tablet orally once daily for 12 weeks.
  OLE Phase: Following Blinded Study Phase, participants willing to enter OLE Phase received open-label cilofexor 100 mg tablet orally once daily for 97.3 weeks.
Period: Blinded Study Phase
Arm/Group | Cilofexor 100 mg | Cilofexor 30 mg | Placebo
Started | 28 | 30 | 13
Completed | 23 | 28 | 12
Not Completed | 5 | 2 | 1
Not completed — Withdrew Consent | 1 | 2 | 1
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Investigator's discretion | 1 | 0 | 0
Period: Open-Label Extension Phase
Arm/Group | Cilofexor 100 mg | Cilofexor 30 mg | Placebo
Started | 23 | 28 | 12
Completed | 5 | 3 | 2
Not Completed | 18 | 25 | 10
Not completed — Study terminated by sponsor | 10 | 12 | 6
Not completed — Adverse Event | 4 | 7 | 3
Not completed — Lack of Efficacy | 3 | 4 | 0
Not completed — Withdrew consent | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Cilofexor 100 mg: Blinded Study Phase: Cilofexor 100 mg tablet + placebo to match cilofexor 30 mg tablet orally once daily for 12 weeks.
  Open Label Extension (OLE) Phase: Following Blinded Study Phase, participants willing to enter OLE phase received open-label cilofexor 100 mg tablet orally once daily for 97.4 weeks.
- Total: Total of all reporting groups
Arm/Group | Cilofexor 100 mg | Cilofexor 30 mg | Placebo | Total
Number analyzed (Participants) | 28 | 30 | 13 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (9.8) | 57 (6.3) | 58 (5.9) | 56 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 12 | 66
  Male | 0 | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race information.
  Participants
    Race: Asian | 2 | 0 | 0 | 2
    Race: Black or African American | 0 | 1 | 0 | 1
    Race: White | 26 | 27 | 13 | 66
    Race: Not Permitted | 0 | 1 | 0 | 1
    Race: Other | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 1 | 1 | 2 | 4
    Ethnicity: Not Hispanic or Latino | 26 | 28 | 11 | 65
    Ethnicity: Not Permitted | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 9 | 3 | 21
  Austria | 4 | 2 | 1 | 7
  United States | 12 | 16 | 7 | 35
  United Kingdom | 3 | 3 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) in the Blinded Study Phase
Time Frame: First dose date up to Week 12 + 30 days
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Blinded Study Phase: Cilofexor 100 mg: Blinded Study Phase: Cilofexor 100 mg tablet + placebo to match cilofexor 30 mg tablet orally once daily for 12 weeks.
- Blinded Study Phase: Cilofexor 30 mg: Blinded Study Phase: Cilofexor 30 mg tablet + placebo to match cilofexor 100 mg tablet orally once daily for 12 weeks.
- Blinded Study Phase: Placebo: Blinded Study Phase: Placebo to match cilofexor 100 mg tablet + placebo to match cilofexor 30 mg tablet orally once daily for 12 weeks.
Arm/Group | Blinded Study Phase: Cilofexor 100 mg | Blinded Study Phase: Cilofexor 30 mg | Blinded Study Phase: Placebo
Number analyzed (Participants) | 28 | 30 | 13
percentage of participants
  TEAEs | 89.3 | 76.7 | 84.6
  TESAEs | 0 | 3.3 | 0

2. Primary Outcome: Percentage of Participants Experiencing TEAEs and TESAEs in the Open-Label Extension (OLE) Phase
Time Frame: First dose date in the OLE phase up to last dose date (Maximum: 97.4 weeks) + 30 days
Population: The OLE Analysis Set included all participants who took at least 1 dose of study drug in the OLE Phase.
Measure: Number; unit: percentage of participants
Groups:
- OLE Phase: From Cilofexor 100 mg: OLE Phase: Following Blinded Study Phase, participants willing to enter OLE Phase received open-label cilofexor 100 mg tablet orally once daily for 97.4 weeks.
- OLE Phase: From Cilofexor 30 mg: OLE Phase: Following Blinded Study Phase, participants willing to enter OLE Phase received open-label cilofexor 100 mg tablet orally once daily for 96.1 weeks.
- OLE Phase: From Placebo: OLE Phase: Following Blinded Study Phase, participants willing to enter OLE Phase received open-label cilofexor 100 mg tablet orally once daily for 97.3 weeks.
Arm/Group | OLE Phase: From Cilofexor 100 mg | OLE Phase: From Cilofexor 30 mg | OLE Phase: From Placebo
Number analyzed (Participants) | 23 | 28 | 12
percentage of participants
  TEAEs | 95.7 | 89.3 | 100.0
  TESAEs | 4.3 | 0 | 0

3. Primary Outcome: Percentage of Participants Who Experienced Graded Laboratory Abnormalities in the Blinded Study Phase
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: First dose date up to Week 12 + 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Study Phase: Cilofexor 100 mg | Blinded Study Phase: Cilofexor 30 mg | Blinded Study Phase: Placebo
Number analyzed (Participants) | 28 | 30 | 13
percentage of participants
  Any Graded Laboratory Abnormality | 85.7 | 86.7 | 92.3
  Grade 4 or above Laboratory Abnormalities | 0 | 3.3 | 0

4. Primary Outcome: Percentage of Participants Who Experienced Graded Laboratory Abnormalities in the OLE Phase
Description: as for outcome 3
Time Frame: First dose date in the OLE phase up to last dose date (Maximum: 97.4 weeks) + 30 days
Population: Participants in the OLE Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- OLE Phase: From Cilofexor 100 mg: OLE Phase: Following Blinded Study Phase, participants in cilofexor 100 mg group, willing to enter OLE Phase received open-label cilofexor 100 mg tablet orally once daily for 97.4 weeks.
- OLE Phase: From Cilofexor 30 mg: OLE Phase: Following Blinded Study Phase, participants in cilofexor 30 mg group, willing to enter OLE Phase received open-label cilofexor 100 mg tablet orally once daily for 96.1 weeks.
- OLE Phase: From Placebo: OLE Phase: Following Blinded Study Phase, participants in placebo group, willing to enter OLE Phase received open-label cilofexor 100 mg tablet orally once daily for 97.3 weeks.
Arm/Group | OLE Phase: From Cilofexor 100 mg | OLE Phase: From Cilofexor 30 mg | OLE Phase: From Placebo
Number analyzed (Participants) | 23 | 28 | 12
percentage of participants
  Any Graded Laboratory Abnormality | 91.3 | 96.4 | 100.0
  Grade 4 or above Laboratory Abnormalities | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Blinded Study Phase: First dose date up to Week 12 + 30 days; Open-label Extension (OLE) Phase: First dose date in the OLE Phase up to last dose date (Maximum: 97.4 weeks) + 30 days
Description: The Safety Analysis Set for Blinded Study phase included all participants who took at least 1 dose of study drug in Blinded Study phase and the OLE Analysis Set included all participants who took at least 1 dose of study drug in OLE phase.
Groups:
- OLE Phase: From Cilofexor 100 mg: OLE Phase: Following Blinded Study Phase, participants in the Cilofexor 100 mg group, willing to enter OLE Phase received open-label cilofexor 100 mg tablet orally once daily for 97.4 weeks.
- OLE Phase: From Cilofexor 30 mg: OLE Phase: Following Blinded Study Phase, participants in the Cilofexor 30 mg group, willing to enter OLE Phase received open-label cilofexor 100 mg tablet orally once daily for 96.1 weeks.
- OLE Phase: From Placebo: OLE Phase: Following Blinded Study Phase, participants in the Placebo group, willing to enter OLE Phase received open-label cilofexor 100 mg tablet orally once daily for 97.3 weeks.
Arm/Group | Blinded Study Phase: Cilofexor 100 mg | Blinded Study Phase: Cilofexor 30 mg | Blinded Study Phase: Placebo | OLE Phase: From Cilofexor 100 mg | OLE Phase: From Cilofexor 30 mg | OLE Phase: From Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30 | 0/13 | 0/23 | 0/28 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/30 | 0/13 | 1/23 | 0/28 | 0/12
Other Adverse Events (participants affected / at risk) | 21/28 | 18/30 | 11/13 | 20/23 | 25/28 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Study Phase: Cilofexor 100 mg (N=28) | Blinded Study Phase: Cilofexor 30 mg (N=30) | Blinded Study Phase: Placebo (N=13) | OLE Phase: From Cilofexor 100 mg (N=23) | OLE Phase: From Cilofexor 30 mg (N=28) | OLE Phase: From Placebo (N=12)
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Study Phase: Cilofexor 100 mg (N=28) | Blinded Study Phase: Cilofexor 30 mg (N=30) | Blinded Study Phase: Placebo (N=13) | OLE Phase: From Cilofexor 100 mg (N=23) | OLE Phase: From Cilofexor 30 mg (N=28) | OLE Phase: From Placebo (N=12)
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 2 | 0 | 0
Dry eye (Eye disorders) | 2 | 0 | 0 | 0 | 2 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 1 | 1 | 6 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 3 | 3 | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 1 | 1
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 5 | 2 | 3 | 3 | 4 | 2
Influenza like illness (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 1 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abscess neck (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1
Carbuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 4 | 5 | 1 | 3 | 4 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 2 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Procedural anxiety (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 3 | 1
Headache (Nervous system disorders) | 4 | 4 | 4 | 2 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 2 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 6 | 3 | 4 | 11 | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT02943447/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT02943447/SAP_001.pdf